CLINICAL TRIAL: NCT05366426
Title: Effect of EMG Biofeedback in Female Patients With Stress Urinary Incontinence
Acronym: 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2022-05-05; First posted 2022-05-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress Urinary Incontinence; EMG biofeedback; Quality of life
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Randomised controlled Trial
Who Masked: Participant, Investigator
Masking Description: The prospective, randomized and controlled interventional study with a three-month follow-up period will be carried out in a single center. Female patients with a clinical diagnosis of stress urinary incontinence will be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Pelvic floor muscle training exercise program will be applied with EMG biofeedback.
  Interventions: Other: EMG biofeedback program:; Other: Pelvic floor muscle training home exercise program:
- Sham Group (Sham Comparator): Pelvic floor muscle training exercise program will be applied with EMG biofeedback as a sham.
  Interventions: Other: Sham EMG biofeededback:; Other: Pelvic floor muscle training home exercise program:
- Control Group (Other): Pelvic floor muscle training program will be applied as home exercise
  Interventions: Other: Pelvic floor muscle training home exercise program:

INTERVENTIONS:
Other: EMG biofeedback program: — Superficial electrodes and EMG-guided biofeedback will be applied to the perineal region 3 days a week for 8 weeks, so that patients can receive visual and auditory feedback during exercise.
  Arms: Experimental group
Other: Sham EMG biofeededback: — 3 days a week for 8 weeks; Surface electrodes will be attached as in the EMG Biofeedback group, but unlike the EMG biofeedback group, they will exercise without any visual and auditory feedback (1).
  Arms: Sham Group
Other: Pelvic floor muscle training home exercise program: — Pelvic floor muscle training home exercise program: A home exercise program was given to all patients who had learned to perform correct pelvic floor muscle contraction with the pre-treatment evaluation. In the home exercise program, patients in three positions (sitting, lying and standing) are required to perform two to three rapid contractions of 15 repetitions in each set, three times a day, followed by slow contractions by keeping the PTC tense for 8-10 seconds, and then give a 10-second rest period after slow contractions. has been told. All 3 groups received PTK exercise program.

SUMMARY:
The aim of this randomized controlled study was to compare the EMG biofeedback method with pelvic floor muscle (PTC) exercises and Sham EMG biofeedback group in women with stress urinary incontinence (SUI) on pelvic floor muscle strength, trunk endurance, subjective perception of improvement, severity of complaints, pad test and quality of life. to determine its effectiveness.

DETAILED DESCRIPTION:
Urogynecological complaints have medical and social aspects that negatively affect quality of life.

are problems. depression, anxiety, low productivity at work, social isolation and associated with sexual dysfunction. Urinary incontinence (UI), which has serious negative effects on people's quality of life, psychological state and physical health, and especially affects older women, stands out as an important public health problem with the prolongation of the average life expectancy. The two most common types of UI in women are stress urinary incontinence (SUI) and urge urinary incontinence (UI). While SUI is the involuntary leakage of urine typically during coughing, sneezing and other physical activities; UUI is defined as urinary incontinence associated with urgency with a sudden and forced need to urinate. The simultaneous presence of SUI and UUI symptoms is defined as mixed urinary incontinence (MUI). Treatment options of SUI, which are divided into conservative and surgical treatment, are conservative treatment options; behavioral therapy (changing lifestyle and dietary habits and bladder training) and PTC rehabilitation (PTK exercises, biofeedback, electrical stimulation, electromagnetic stimulation, neuromodulation and vaginal issues). With PTK exercises, it is aimed to work the levator ani muscle group. These exercises are described as contractions and relaxation periods lasting 10 seconds. It is recommended to be applied in 3 different positions while lying, sitting and standing. Increasing the number of contractions gradually and reaching 60 repetitions per day is targeted in the treatment (1).

One of the ways to teach PTK exercises is "biofeedback" (BF). This method provides visual and auditory feedback while teaching the correct contraction of the muscles (2). Since it is an active method, it is thought that the increase in PTK power is higher. Superficial or internal electrodes can be used (3). The investigators will use surface electrodes in our project. In a recent meta-analysis in the literature (4); In the current meta-analysis on the effectiveness of EMG biofeedback in patients with SUI, it was reported that pelvic floor muscle training combined with EMG-BF achieved better results than pelvic floor muscle training alone in the management of SUI, but randomized studies are still needed to confirm the results.

To determine the effectiveness of EMG biofeedback method on pelvic floor muscle strength, severity of complaints, pad test and quality of life in women with stress urinary incontinence (SUI) by comparing them with pelvic floor muscle (PTK) exercises and Sham EMG biofeedback group.

In our project, the investigators will be able to determine whether the EMG biofeedback exercise performed with the device is really superior to the exercise performed by the patient himself, using the Sham group. Thus, the results of our project; It will provide scientific data for teaching patients about pelvic floor muscle training in the clinic and for use in urinary rehabilitation of SUI patients.

ELIGIBILITY:
Inclusion Criteria:

1.30-65 years old women clinical diagnoses of Urinary Incontinence 2. Clinical diagnoses of Stress Urinary Incontinence (SUI) or Mixt Urinary Incontinence (MUI) with a dominant Stress Urinary Incontinence component 3.Must be have not received treatment with any physical therapy modality in the last 3 months 4.Must be urinary incontinence severity of at least 5 points on Visual Analog Scale 5.Must be able to signed the informed consent form

Exclusion Criteria:

1. Severe systemic disease that prevents exercise (Cardiovascular disease, COPD, CVO and/or cancer)
2. Pure urge or MUI with a dominant urge component
3. Plan to change or change medical treatment within the last 3 months due to UUI
4. Visual, auditory, or cognitive deficits that are not suitable for treatment requirements
5. High-intensity sports activities for at least half an hour, at least 2 times a week

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients
Enrollment: 60 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-04-07 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
International Incontinence Inquiry Form ICIQ-SF | 0 (baseline)
  International Incontinence Inquiry Form ICIQ-SF Avery et al. and it was reported that the sensitivity, reliability and validity of the scale were high (1). The scale is available in four dimensions. In the first dimension, the frequency of urinary incontinence, the amount of urinary incontinence in the second dimension, the effect of urinary incontinence on daily life in the third dimension, and the conditions that cause urinary incontinence in the fourth dimension are questioned. It was validated in Turkish in 2004 and started to be used in our country.
International Incontinence Inquiry Form ICIQ-SF | 8th week (after treatment)
  International Incontinence Inquiry Form ICIQ-SF Avery et al. and it was reported that the sensitivity, reliability and validity of the scale were high (1). The scale is available in four dimensions. In the first dimension, the frequency of urinary incontinence, the amount of urinary incontinence in the second dimension, the effect of urinary incontinence on daily life in the third dimension, and the conditions that cause urinary incontinence in the fourth dimension are questioned. It was validated in Turkish in 2004 and started to be used in our country.
International Incontinence Inquiry Form ICIQ-SF | 20th week (3 months after treatment)
  International Incontinence Inquiry Form ICIQ-SF Avery et al. and it was reported that the sensitivity, reliability and validity of the scale were high (1). The scale is available in four dimensions. In the first dimension, the frequency of urinary incontinence, the amount of urinary incontinence in the second dimension, the effect of urinary incontinence on daily life in the third dimension, and the conditions that cause urinary incontinence in the fourth dimension are questioned. It was validated in Turkish in 2004 and started to be used in our country.
Pad test; | 0 (baseline)
  Pad test; It is one of the objective tests showing the presence and degree of UI. In the one-hour pad test standardized by ICS, the patient is asked to use a pad of known weight for one hour following 500 mL of non-sodium oral hydration for 15 minutes without urinating. During this period, 30 patients walking, going up and down stairs, sitting up 10 times, coughing 10 times, running for 1 minute, bending down 5 times and washing hands for 1 minute. The weight difference measured on the pad at the end of 1 hour is considered to indicate the amount of urine that has escaped. This amount; If it is less than 1 gram, it is definitely dry, if it is between 2-10 grams, it is considered as mild moderate urinary incontinence, between 10-50 grams as severe urinary incontinence, and over 50 grams as very severe urinary incontinence. To increase the reliability of the test, the duration of the test can be extended from 2 hours to 48 hours.
Pad test; | 8th week (after treatment)
  Pad test; It is one of the objective tests showing the presence and degree of UI. In the one-hour pad test standardized by ICS, the patient is asked to use a pad of known weight for one hour following 500 mL of non-sodium oral hydration for 15 minutes without urinating. During this period, 30 patients walking, going up and down stairs, sitting up 10 times, coughing 10 times, running for 1 minute, bending down 5 times and washing hands for 1 minute. The weight difference measured on the pad at the end of 1 hour is considered to indicate the amount of urine that has escaped. This amount; If it is less than 1 gram, it is definitely dry, if it is between 2-10 grams, it is considered as mild moderate urinary incontinence, between 10-50 grams as severe urinary incontinence, and over 50 grams as very severe urinary incontinence. To increase the reliability of the test, the duration of the test can be extended from 2 hours to 48 hours.
Pad test; | 20th week (3 months after treatment)
  Pad test; It is one of the objective tests showing the presence and degree of UI. In the one-hour pad test standardized by ICS, the patient is asked to use a pad of known weight for one hour following 500 mL of non-sodium oral hydration for 15 minutes without urinating. During this period, 30 patients walking, going up and down stairs, sitting up 10 times, coughing 10 times, running for 1 minute, bending down 5 times and washing hands for 1 minute. The weight difference measured on the pad at the end of 1 hour is considered to indicate the amount of urine that has escaped. This amount; If it is less than 1 gram, it is definitely dry, if it is between 2-10 grams, it is considered as mild moderate urinary incontinence, between 10-50 grams as severe urinary incontinence, and over 50 grams as very severe urinary incontinence. To increase the reliability of the test, the duration of the test can be extended from 2 hours to 48 hours.
The King's Health Questionnaire | 0 (baseline)
  The King's Health Questionnaire (KSA) is a two-part questionnaire that includes 32 items and is frequently used to evaluate the quality of life of patients with incontinence. In addition to two single-item questions such as general health status and impact on quality of life, it includes 7 sub-headings consisting of multiple items. These include: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, sleep and energy disturbances associated with incontinence, and severity measures for incontinence. The second part is the 11-item Symptom Severity Scale, which assesses the presence and severity of urinary symptoms. The score of the Symptom Severity Scale ranges from 0 (best) to 30 (worst). Scores for other KSA domains range from 0 (best) to -100 (worst). Turkish validity and reliability was established (3).
The King's Health Questionnaire | 8th week (after treatment)
  The King's Health Questionnaire (KSA) is a two-part questionnaire that includes 32 items and is frequently used to evaluate the quality of life of patients with incontinence. In addition to two single-item questions such as general health status and impact on quality of life, it includes 7 sub-headings consisting of multiple items. These include: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, sleep and energy disturbances associated with incontinence, and severity measures for incontinence. The second part is the 11-item Symptom Severity Scale, which assesses the presence and severity of urinary symptoms. The score of the Symptom Severity Scale ranges from 0 (best) to 30 (worst). Scores for other KSA domains range from 0 (best) to -100 (worst). Turkish validity and reliability was established (3).
The King's Health Questionnaire | 20th week (3 months after treatment)
  The King's Health Questionnaire (KSA) is a two-part questionnaire that includes 32 items and is frequently used to evaluate the quality of life of patients with incontinence. In addition to two single-item questions such as general health status and impact on quality of life, it includes 7 sub-headings consisting of multiple items. These include: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, sleep and energy disturbances associated with incontinence, and severity measures for incontinence. The second part is the 11-item Symptom Severity Scale, which assesses the presence and severity of urinary symptoms. The score of the Symptom Severity Scale ranges from 0 (best) to 30 (worst). Scores for other KSA domains range from 0 (best) to -100 (worst). Turkish validity and reliability was established (3).

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asisst Prof, Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kırşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terlikowski R, Dobrzycka B, Kinalski M, Kuryliszyn-Moskal A, Terlikowski SJ. Transvaginal electrical stimulation with surface-EMG biofeedback in managing stress urinary incontinence in women of premenopausal age: a double-blind, placebo-controlled, randomized clinical trial. Int Urogynecol J. 2013 Oct;24(10):1631-8. doi: 10.1007/s00192-013-2071-5. Epub 2013 Feb 27. PMID 23443345
- [Background] Wu X, Zheng X, Yi X, Lai P, Lan Y. Electromyographic Biofeedback for Stress Urinary Incontinence or Pelvic Floor Dysfunction in Women: A Systematic Review and Meta-Analysis. Adv Ther. 2021 Aug;38(8):4163-4177. doi: 10.1007/s12325-021-01831-6. Epub 2021 Jun 27. PMID 34176082